CLINICAL TRIAL: NCT04249830
Title: Allogeneic Hematopoietic Stem Cell Transplantation From an HLA-partially Matched Related or Unrelated Donor After TCR αβ+T Cells/CD19+ B Cell Depletion in Children and Young Adults Affected by Malignant or Non-Malignant Hematological Disorders
Brief Title: Stem Cell Transplant From Donors After Alpha Beta Cell Depletion in Children and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alice Bertaina (Other)
Responsible Party: Sponsor-Investigator, Alice Bertaina, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-53822; BMT 361 - Alpha Beta IDE (Other: Stanford School of Medicine)
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Stem Cell Transplant -Malignant (Experimental): The participant with a malignancy will undergo a stem cell transplant using donor cells that have been manipulated through an investigational device. Participants will be followed for outcomes for two years.
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS TCR α/β Reagent Kit and CliniMACS CD19
- Stem Cell Transplant - Non-Malignant (Experimental): The participant with a non-malignant disease will undergo a stem cell transplant using donor cells that have been manipulated through an investigational device. Participants will be followed for outcomes for two years.
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS TCR α/β Reagent Kit and CliniMACS CD19
- Stem Cell Transplant - Compassionate (Other): Patients with malignant or non-malignant disorders who do not qualify for experimental arms but who may still benefit from participation in this study may be enrolled in this arm.
  Interventions: Biological: Allogeneic Stem Cell Transplant; Device: CliniMACS TCR α/β Reagent Kit and CliniMACS CD19

INTERVENTIONS:
Biological: Allogeneic Stem Cell Transplant — The allogeneic stem cell transplant involves transferring the stem cells from a healthy person (donor) to the participant via infusion.
Device: CliniMACS TCR α/β Reagent Kit and CliniMACS CD19 — The CliniMACS™system can be used to selectively enrich or reduce specific cell populations based on the magnetic cell selection (MACS) technology developed by Miltenyi Biotec. Cell mixtures can be separated in a magnetic field using one or more immunomagnetic- labeled antibodies specific for the cell types of interest (e.g.TCR αβ+ T cells and CD19+ B cells from HPC(A) products).

SUMMARY:
The purpose of the CliniMACS® TCRαβ-Biotin System and CliniMACS® CD19 is to improve the safety and efficacy of allogeneic HLA-partially matched related or unrelated donors HSCT when no matched donors are available, to treat malignant and nonmalignant disorders for which HSCT is the recommended best available therapy. Initially this device will be used in a single-center, open-label, single-arm, phase II clinical trial to evaluate the efficacy of haploidentical PBSC grafts depleted of TCRα/β+ and CD19+ cells using the CliniMACS® TCRαβ/CD19 System in children and adults with hematological and non-hematological malignancies.

ELIGIBILITY:
Inclusion Criteria for Cohort M and Cohort NM:

1. Age < 60 years and > 1 month;
2. Life expectancy > 10 weeks;
3. Patients deemed eligible for allogeneic HSCT per institutional guidelines;
4. Patients with life-threatening hematological malignancies and non-malignant disorders that could benefit from HSCT;

   a. For malignant patients: i. High-risk acute lymphoblastic leukemia (ALL) in 1st complete remission (CR), ALL in 2nd CR; or ii. High-risk acute myeloid leukemia (AML) in 1st CR, AML in 2nd CR; or iii. Childhood Myelodysplastic Syndrome (MDS) with low blasts (cMDS-LB) or Childhood MDS with increased blasts (cMDS-IB); or iv. Juvenile myelomonocytic leukemia (JMML); or v. Mixed-phenotype acute leukemia (MPAL); or vi. Non-Hodgkin lymphomas in 2nd CR; or vii. Other hematologic malignancies in 1st or 2nd CR eligible for stem cell transplantation per institutional standard b. Patients with non-malignant disorders receiving first HSCT: i. using mis-matched donors, due to the absence of suitable HLA identical sibling or HLA phenotypically identical relative; or ii. whose disease put them at increased risk of graft rejection or GvHD (e.g., Fanconi Anemia, STAT1 gain of function) and therefore can benefit from receiving alpha beta depleted HSCT using as a donor either an HLA identical sibling or an HLA phenotypically identical (10/10 matched) donor;
5. A minimum genotypic identical match of 5/10 is required;
6. The donor and recipient must be identical, as determined by high resolution typing, in at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-C, HLA-DQB1 and HLA-DRB1;
7. Lansky/Karnofsky score > 50; the Karnofsky Scale will be used in subjects ≥ 16 years of age, and the Lansky Scale will be used for those < 16 years of age.
8. All subjects ≥ 18 years of age must be able to give informed consent or adults lacking capacity to consent must have a legally authorized representative (LAR) available to provide consent. For subjects <18 years old their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age appropriate discussion and written assent will be obtained for those > 7 years of age, when appropriate
9. Male and female subjects of childbearing potential must agree to use an effective means of birth control to avoid pregnancy throughout the transplant procedure, while on immunosuppression, and if the subject experiences any chronic GvHD.

Exclusion Criteria for Cohort M and Cohort NM:

1. Pregnant or lactating females;
2. Has received a prior allogenic HSCT;
3. Secondary MDS or AML or treatment related MDS or AML;
4. Dysfunction of liver (ALT/AST > 10 times upper normal value, or direct bilirubin > 3 times upper normal value),
5. Serum creatinine > 1.5 times ULN (for patients not on dialysis) or unmanageable dysfunction of renal function while undergoing dialysis (for patients on dialysis);
6. Severe cardiovascular disease (congestive heart failure or left ventricular ejection fraction < 30%);
7. Current active infectious disease (including positive HIV serology or viral RNA);
8. Serious concurrent uncontrolled medical disorders;
9. Lack of patient's/parents'/guardian's informed consent;
10. Any severe concurrent disease which, in the judgement of the PI, would place the patient at increased risk during participation in the study.

Ages: 1 Month to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with grade II-IV acute GvHD after HSCT | Through Day 100 after HSCT

SECONDARY OUTCOMES:
Leukemia-free survival after HSCT | 1 and 2 years after HSCT
  Leukemia-free survival defined as the time of enrollment to disease relapse or death from any cause.
Number of participants with secondary graft failure at after HSCT | 1 and 2 year after HSCT
Number of participants with grade III-IV acute GvHD after HSCT | Through Day 100 after HSCT
Incidence rate of primary graft failure after HSCT | Day 42 after HSCT
Incidence of moderate and severe chronic GvHD after HSCT | 1 year after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: David Shyr, MD, Principal Investigator — Clinical Associate Professor, Pediatrics, Stem Cell Transplantation
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No